CLINICAL TRIAL: NCT05636995
Title: HyperAldosteronism in Pregnancy Predicted Impacts
Brief Title: HyperAldosteronism in Pregnancy Predicted Impacts (H.A.P.P.I. Trial)
Status: Active, not recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Nadine Sauvé, Principal investigator, Université de Sherbrooke
Other Study IDs: MP-31-2023-4857
Record Dates: First submitted 2022-10-25; First posted 2022-12-05 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Primary Hyperaldosteronism; Hypertensive Disorder of Pregnancy
Keywords: Pregnancy Outcome; Prevalence
MeSH Terms: conditions — Hyperaldosteronism; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary Hyperaldosteronism Diagnosed Women: Post-partum women who had a hypertensive disorder of pregnancy and a screened primary hyperaldosteronism (positive aldosterone/renin ratio).
  Interventions: Diagnostic Test: Aldosterone/Renin Ratio
- Control Women: Post-partum women who had a hypertensive disorder of pregnancy without underlying primary hyperaldosteronism (negative aldosterone/renin ratio)
  Interventions: Diagnostic Test: Aldosterone/Renin Ratio

INTERVENTIONS:
Diagnostic Test: Aldosterone/Renin Ratio — Blood sample collected to measure the aldosterone/renin ratio for the primary hyperaldosteronism screening.

SUMMARY:
Primary hyperaldosteronism confers a higher risk of cardiovascular complications compared to essential hypertension. Preliminary data is controversial in regards of excessive maternal fetal and neonatal excessive risks in pregnancy.

This study aims at establishing the prevalence of PHA in an population with a recent episode of hypertensive disorder of pregnancy (HDP). The goal is to determine if a universal screening for PHA after a HDP is worthed. The investigators also wish to evaluate the complication rate in pregnant women with PHA compared to women without PHA.

This is a prospective cohort study where all eligible women will be screened for PHA after a HDP episode in the last pregnancy. We will then compare PHA women to non PHA women according to pregnancy complications.

DETAILED DESCRIPTION:
This is a pilot study to evaluate feasibility and proof of concept. This is a prospective multicenter cohort study. Two university centers will participate (Sherbrooke and Montreal).

Participants will be recruited from post-partum Obstetric Medicine clinic in two tertiary care centers. They will be included if they presented a hypertensive disorder of preganncy (HDP) in their last pregnacy (from 4 weeks to 24 months after delivery). Women with pheochromocytoma, Cushing syndrome, secondary hyperaldosteronism, and those who are currently pregnant will be excluded.

All participants will be screened for PHA (with an aldosterone/renin ratio) and if the screening test is positive, they will be referred to a specialist to confirm the diagnosis.

Data will be collected from the participants and their babies' charts. Demographic data, obstetrical data, delivery data, maternal/fetal/neonatal complications, and diagnostic of PHA data will be collected.

A convenient sample size of 200 women will be used. If the prevalence of HPA is 5% or more, this would justify a larger study.

Primary outcome: establish the prevalence of PHA in women with a hypertensive disorders of pregnancy in last pregancy.

Secondary outcome include:

1. to compare maternal, fetal and neonatal outcomes among women diagnosed with primary hyperaldosteronism (PHA) and pregnant women without PHA.
2. to establish the prevalence of PHA for each sub-type of hypertensive disorder of pregnancy
3. to compare maternal, fetal and neonatal outcomes among women diagnosed with primary hyperaldosteronism (PHA) before pregnancy and pregnant women diagnosed with PHA after pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Between 4 and 24 weeks post-partum women who had a hypertensive disorder during their latest pregnancy.

Exclusion Criteria:

* Ongoing pregnancy
* Diagnosed pheochromocytoma
* Diagnosed Cushing syndrome
* Diagnosed secondary hyperaldosteronism

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-partum women who are followed in a specialized post-partum clinic in Montreal or Sherbrooke (Qc, Canada) for their hypertensive disorder during their latest pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary hyperaldosteronism (PHA) prevalence in pregnant women with hypertensive disorders of pregnancy. | Screening done between 4 and 24 weeks post-partum
  Prevalence of PHA in women with a hypertensive disorder of pregnancy in last pregnancy

SECONDARY OUTCOMES:
Maternal and fetal impacts of PHA on hypertensive disorders of pregnancy | During last pregnancy and 6 weeks postpartum
  Comparison of the prevalence of each pre-specified complications (obstetrical, maternal, fetal, neonatal) between the PHA group and the non-PHA group.
Prevalence of PHA for each hypertensive disorder of pregnancy | During last pregnancy and 6 weeks postpartum
  Comparison of the prevalence of each HDP subtype (i.e. chronic hypertension, gestational hypertension, pre-eclampsia)
Impact of the timing of PHA on hypertensive disorders of pregnancy | During last pregnancy and 6 weeks postpartum
  Comparison between pregnancy outcomes for PHA diagnosed before the pregnancy with those diagnosed in post-partum

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Sauvé, MD, Principal Investigator — Université de Sherbrooke
Locations (2):
- Canada (2):
  - Centre Hopitalier Universiatire de Sherbrooke, Sherbrooke, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alam S, Kandasamy D, Goyal A, Vishnubhatla S, Singh S, Karthikeyan G, Khadgawat R. High prevalence and a long delay in the diagnosis of primary aldosteronism among patients with young-onset hypertension. Clin Endocrinol (Oxf). 2021 Jun;94(6):895-903. doi: 10.1111/cen.14409. Epub 2021 Feb 22. PMID 33393127
- [Background] Magee LA, Pels A, Helewa M, Rey E, von Dadelszen P; Canadian Hypertensive Disorders of Pregnancy Working Group. Diagnosis, evaluation, and management of the hypertensive disorders of pregnancy: executive summary. J Obstet Gynaecol Can. 2014 May;36(5):416-41. doi: 10.1016/s1701-2163(15)30588-0. English, French. PMID 24927294
- [Background] Turner K, Hameed AB. Hypertensive Disorders in Pregnancy Current Practice Review. Curr Hypertens Rev. 2017;13(2):80-88. doi: 10.2174/1573402113666170529110024. PMID 28554307
- [Background] Umesawa M, Kobashi G. Epidemiology of hypertensive disorders in pregnancy: prevalence, risk factors, predictors and prognosis. Hypertens Res. 2017 Mar;40(3):213-220. doi: 10.1038/hr.2016.126. Epub 2016 Sep 29. PMID 27682655
- [Background] Landau E, Amar L. Primary aldosteronism and pregnancy. Ann Endocrinol (Paris). 2016 Jun;77(2):148-60. doi: 10.1016/j.ando.2016.04.009. Epub 2016 May 6. PMID 27156905
- [Background] Downie E, Shanmugalingam R, Hennessy A, Makris A. Assessment and Management of Primary Aldosteronism in Pregnancy: A Case-Control Study. J Clin Endocrinol Metab. 2022 Jul 14;107(8):e3152-e3158. doi: 10.1210/clinem/dgac311. PMID 35569086
- [Background] Escher G. Hyperaldosteronism in pregnancy. Ther Adv Cardiovasc Dis. 2009 Apr;3(2):123-32. doi: 10.1177/1753944708100180. Epub 2009 Jan 26. PMID 19171690